CLINICAL TRIAL: NCT06877091
Title: Nutritional Status and Intake in Patients With Non-cystic Fibrosis Bronchiectasis (NCFB) - a Cross Sectional Study
Brief Title: Nutritional Status and Intake in Patients With Non-cystic Fibrosis Bronchiectasis (NCFB)
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Collaborators: The Leeds Teaching Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Professor Daniel G Peckham, Professor, University of Leeds
Other Study IDs: Version 1
Record Dates: First submitted 2025-03-06; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Non Cystic Fibrosis Bronchiectasis
Keywords: Nutritional status; Dietary Intake; NCFB

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Regional cohort of individuals living with Non-Cystic Fibrosis Bronchiectasis

SUMMARY:
The aim of this study was to characterise nutritional status and dietary intake in a population of individuals living with bronchiectasis from a regional clinic. Participants underwent usual assessment as per their standard pathway of care and in addition, body composition through skinfold measures, Handgrip strength and information on dietary intake over 3 days via 24 hour multiple pass recalls was also collected. This was to establish baseline measures and knowledge in support of understanding the impact of nutritional status within this group.

ELIGIBILITY:
Inclusion Criteria:

* People who have a confirmed diagnosis of NCFB
* people with NCFB who are clinically stable (not requiring acute admission to hospital)
* people who attend the regional clinic

Exclusion Criteria:

* People who are pregnant
* people with existing comorbidities such as malignancy

Ages: 17 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Those who attend the Leeds Regional Bronchiectasis Clinic
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Lung Function (FEV1 ) | At point of recruitment
  Collect spirometry data that is measured as part of clinical care
Lung Function ( FVC) | At point of recruitment
  Collect spirometry data that is measured as part of clinical care
Height (m) | At point of recruitment
  Height will be taken to enable measurement of BMI
Weight (kg) | At point of recruitment
  Weight will be taken to provide unit to calculate BMI (kg/m2)
BMI (kg/m2) | At point of recruitment
  Collection of standard data (weight and height) from usual care pathway

SECONDARY OUTCOMES:
Handgrip Dynamometry (kg/f) | At point of recruitment
  Collection of hand grip strength to establish a mean value
Tricep Skinfold measurement (mm) | At point of recruitment
  To measure triceps skinfold to determine estimated fat mass
Dietary intake checklist | At point of recruitment
  To collect 3 separate 24 hour recalls over multiple days to establish mean reported intakes.

CONTACTS AND LOCATIONS:
Locations (1):
- Leeds Teaching Hospitals Trust, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
This study was undertaken in 2017